CLINICAL TRIAL: NCT06074653
Title: Comparative Effects of Mulligan Bent Leg Raise and Contract Relax Technique on Hamstring Flexibility in Office Workers
Brief Title: Effects of Mulligans BLR and CR on Hamstrings Flexibility in Office Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/0164Amna Pervaiz
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Muscle Tightness
Keywords: hamstring tightness; contract relax; mulligan bent leg raise; office worker

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group A (Experimental): Subjects will receive 8 sessions of Mulligan Bent Leg Raise technique on dominant side
  Interventions: Other: Mulligan Bent Leg Raise technique
- Experimental group B (Experimental): Subjects will receive 8 sessions of PNF Contract Relax technique on dominant side
  Interventions: Other: PNF Contract Relax technique

INTERVENTIONS:
Other: Mulligan Bent Leg Raise technique — Treatment session will be conducted for 2 days a week for 4 weeks consecutively. In first week only 20 minutes session will be given to each group. Home exercise plan is also given.Pre and post intervention measurements will be taken at 2nd and 4th week. Both dominant and non-dominant legs will be checked
  Arms: Experimental group A
Other: PNF Contract Relax technique — Treatment session will be conducted for 2 days a week for 4 weeks consecutively. In first week only 20 minutes session will be given to each group. Home exercise plan is also given. Pre and post intervention measurements will be taken at 2nd and 4th week. Both dominant and non-dominant legs will be checked
  Arms: Experimental group B

SUMMARY:
The aim of this research is to compare the effect of mulligan bent leg raise and contract relax technique on hamstring flexibility in office workers with sedentary life styles.

DETAILED DESCRIPTION:
Flexibility is regarded as a crucial component of typical biomechanical operation. A tight hamstring increases the risk of frequent impairment to the associated musculature and bony structure. Hamstring muscles are associated with lumbar spine, pelvic and lower limb movement disorders and have been connected to low back discomfort and abnormal gait pattern. It has been observed that long sitting and sedentary life style is directly related to reduce the hamstrings flexibility, so the persons with tight hamstrings are more prone to develop musculoskeletal disorders if not addressed properly. Previous research has shown that contract relaxation and Mulligan's bent leg are both useful for increasing hamstring flexibility. But there hasn't been much research comparing the two methods, Mulligan bent leg lift and contract relax, for hamstring muscle stiffness in middle age office employees; instead, it was done in young people and athletes. Hence, the aim of present work is to study and compare the effectiveness of contract relax and Mulligan bent leg raise in middle age office workers with long sitting hours having hamstring tightness

ELIGIBILITY:
Inclusion Criteria:

* Middle age men and women (30 to 45 years)
* Working/ sitting hours ≥ 36 hours per week.
* Real estate and IT office workers.
* Participant with positive Active Knee Extension Test: A lag of 20degrees is considered normal from full extension, anything less than 20degrees is considered as hamstrings tightness

Exclusion Criteria:

* History of knee and hip injury
* Neurological impairment
* Other orthopedic conditions i.e., hip fracture, THR, TKR etc
* Fracture of lower limb

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Active Knee Extension Test | 4 weeks
  AKE test with goniometry will be used to evaluate hamstring tightness. Goniometer was used to measure the popliteal angle. When popliteal angle becomes greater than 20 degrees then it's considered as Hamstring tightness. "change will be measured from baseline to 4 weeks"
Lower Extremity Functional Mobility Scale | 4 weeks
  The Lower Extremity Functional Mobility Scale will tell us about activities done by a healthy individual using their lower limbs. The test-retest reliability is excellent ranging between 0.855 and 0.99. "Change will be measured from baseline to 4 weeks"

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Ashraf, TDPT, Principal Investigator — Riphah International University; Amna Pervaiz, MS OMPT*, Principal Investigator — Riphah International University
Locations (1):
- Bari Builders and IT path limited, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No